CLINICAL TRIAL: NCT04894344
Title: Education to Decrease in Sodium Intake in University Students Evaluated With 24 Hour Urinary Sodium Excretion: Randomized Controlled Trial
Brief Title: Education to Decrease in Sodium Intake Evaluated With 24 Hour Urinary Sodium Excretion (RCT)
Acronym: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autonoma de Baja California (Other)
Responsible Party: Principal Investigator, Naysin Yaheko Pardo Buitimea, Professor, Universidad Autonoma de Baja California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ArchiveBioethicsCommittee/245
Record Dates: First submitted 2020-12-27; First posted 2021-05-20 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Hypertension; Overweight or Obesity; Diabetes Mellitus, Type 2
Keywords: Collections, Urine Specimen; Diets, Healthy; Lifestyle; Mentoring; Planning,Health; Sodium,Dietary; Females; Males
MeSH Terms: conditions — Hypertension; Overweight; Obesity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Two groups will be formed, the intervention group and the control group. Participants shall be randomly assigned to one of the two groups. Each patient group receives a single treatment simultaneously Urine measured 24 hours before and after the procedure as well as other variables of interest. The duration of the intervention will be 4 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Educational program (Experimental): Participants will be randomly assigned. Intervention Group: 57 participants Each participant will receive the same educational information throughout the study, each week a newsletter will be provided with recommendations and information that teaches them to choose low-sodium foods for 4 weeks.
  Urine samples of 24 h before and after the Intervention will be analyzed.
  Interventions: Behavioral: Education group
- Control group (No Intervention): Participants will be randomly assigned. Control group:57 participants Follow-up for 4 weeks. Urine samples of 24 h before and after the educational program will be analyzed.

INTERVENTIONS:
Behavioral: Education group — Is taught to choose low-sodium foods
  Arms: Educational program

SUMMARY:
WHO identifies as an important risk factor and potentially modifiable to high sodium intake (>2g/day 5g salt/day). Also, an insufficient consumption of potassium ( 3.5 g/day).Therefore, the results of this research could be the regional basis that is required to generate evidence, that designs strategies and recommendations for the prevention or decrease in the progression of high blood pressure. The reduction in the consumption of salt in the diet could comply with the recommendations established by international agencies. In addition, to favor the beginning of lifestyle changes, as well as other modifications that will have a positive impact on health.In population highly vulnerable to the campaigns of large industries that favor the consumption of processed food.

However, it is unknown what is the effect of reducing foods high in sodium in populations in different regions of Mexico, estimated by 24 hour urine sodium excretion.

Therefore, the present study aims to answer the following questions:

What impact does an intervention aimed at the decrease in sodium intake, in young university students on blood pressure and the quantification of the excretion of sodium and urinary potassium of 24h? What is the association between body mass index, blood pressure and sodium reduction in the intervention vs control group? To assess the impact of an intervention aimed at reducing sodium intake through education as general recommendations for limiting specific foods high in sodium, in university students on blood pressure and quantification of urinary sodium and potassium excretion of 24h.

Specific objectives Assess sodium intake between the intervention group and the control group by estimating 24-hour urinary sodium excretion.

secundary objectives Evaluate the effect between the intervention group and the control group on blood pressure.

To assess the levels of potassium excretion in the intervention and control groups.

To evaluate the association between body mass index, blood pressure and sodium reduction in the intervention and control groups.

DETAILED DESCRIPTION:
According to reports from the World Health Organization (WHO) in 2015, the prevalence of hypertension in the world is 1.13 billion people, representing 1 in 4 men and 1 in 5 women (WHO, 2019). In the Americas, every year 1.6 million people die from cardiovascular disease and it has been reported that 20-40% of the adult population suffer hypertension, representing 250 million people affected.

High salt intake (NaCl) is considered an essential risk factor in the development and progression of hypertension.In addition, several studies indicate that sodium in the diet is directly associated with blood pressure.Deleterious effects of high sodium intake associated with endothelial damage have also been reported in normotensive individuals independent of high blood pressure , reduced endothelial function and microvascular reactivity due to oxidative stress.Likewise, a decrease in the nitric oxide of the endothelium has been described that precedes the development of atherosclerotic plaques, which is known through a mechanism where nitric oxide inhibits platelet aggregation, the adhesion of platelets to collagen fibers and other adhesive proteins, as well as the stimulation of adipocyte hypertrophy by increasing the enzymatic activity of leptin and lipogenic enzymes .With type 2 diabetes mellitus (DM2) and increased insulin resistance through hemodynamic changes in the kidneys by sustained sodium reabsorption.In addition, high salt intake has also been associated with kidney disease, osteoporosis, kidney stone formation and stomach cancer.Recently, as a potential modulator of inflammatory and autoimmune diseases through direct and indirect mechanisms of cellular immunity.Therefore, international organizations recommend decreasing sodium intake in the diet. The WHO recommends that sodium intake be 2000 mg/d (equivalent to 5g of salt) and potassium intake 3.5 g/d in adults, to prevent chronic diseases such as hypertension, risk of heart disease and stroke.

Methodology Study design: a randomized controlled, parallel-group, prospective trial was conducted.

Sample: n= 114, undergraduate students from the Autonomous University of Baja California.

For the sample size of the comparison of two repeated averages in two different groups of participants.Public-Public Software was used for its calculationGRANMO developed by the URLEC Consortium of the research groups on Cardiovascular Risk and Nutrition and on Epidemiology and Cardiovascular Genetics of the IMIM-Hospital del Mar Research Program on Inflammatory and Cardiovascular Processes.

Variables Weight: To be measured with a scale brand TANITA Digital Body Fat Scale for Composition Monitor. Model BC-730F FitScan, (Tokyo, Japan), accurate to 0.1 Kg. Participants will be weighed with light clothing and without shoes.

Size: The size shall be measured without shoes and by the use of a SECA 213 (Hamburg, Germany) statistic, accurate to 0.1cm.

Body Mass Index (BMI): To be calculated according to the following formula: BMI= Weight (kg)/Size2 (cm). And it will be classified according to the criteria established by the WHO in: normal weight (18.5 to 25.0 kg/m2), overweight (25 to 30 kg/m2) and obesity ( 30 kg/m2).

Blood Pressure (BP): slope of the equipment (an automatic digital tensiometer validated for example OMRON will be used, according to the protocol for determining the sodium concentration.

Urinary excretion of sodium and potassium of 24h: It will be calculated by the method of selective electrons of ions in the Specialized Clinical Laboratory of Hematology and Transfusion Unit.

Intervention group Low sodium diet: Restriction of foods with high sodium content through educational newsletters once a week for 4 weeks control group Usual diet Age: 18- 30 years Gender: Male will be coded as 1, and female as 2 at the time of being captured in the database.

Weight: stage diagnosis according to body mass index, categories of normopeso, overweight or obesity according to the WHO.

Diagnosis of blood pressure: according to The eighth Joint National Committee guidelines (JNC 8) published in 2014.

Statistical Analysis: a sample size per group was calculated, with a statistical power of 80% to two tails, with a p= 0.05 to detect a difference of 1000 mg of sodium.A descriptive analysis shall be made of each of the variables expressed according to their level of measurement (averages or medians) with their respective dispersion measurement.

body mass index will be analyzed by category and sex for categorical data with the square Pearson's chi-squared test.

Correlation and simple linear regression shall be applied for body mass index, blood pressure and 24 hour sodium urinary excretion prior to the intervention.

The Student t test will be applied for related samples. Assumptions will be sought for parametric statistical analysis and the corresponding statistical test will be applied if the assumptions are met.The student t-test shall be applied for independent samples and mean differences in the intervention vs control group shall be analysed for 24-hour urinary sodium excretion data.The Kolmogorov-Smirnov test will be applied to see if there is a normal distribution.The Levene statistic shall be applied to assess homoscedasticityThe ANOVA test of a factor to analyze mean difference in the intervention group vs control group, in urinary sodium excretion by sex, will be applied.FACTORIAL ANOVA shall be applied to analyse mean difference in the intervention group vs control group in urinary sodium excretion (the same for potassium excretion) with the BMI categories, sex, for the categories of a low sodium diet (less 2000 mg of Na) and the categories of a standard sodium diet( greater than 3500 mg Na).

Procedure:

The study was submitted for authorization to the graduate committee of the Doctorate in Nutrition and Behavioral Sciences and to the ethics committee of the University Autonomous of Baja California.

Explanation of study purpose to participants and signature of informed consent. Details of how to collect the sample shall be given and the day and time of delivery indicated. A plastic canister with 24h urine collection capacity will be provided.

Blood pressure determination: Participants will be advised not to exercise, eat, drink, or smoke 30 minutes before taking their blood pressure. Before measuring the blood pressure, the participant will be asked to sit in a comfortable and quiet place for at least five minutes, with his back supported and without crossing his legs. When asking questions about behavior and personal medical history, just before taking the measurements, the participant should rest at least five minutes before starting the blood pressure test.

WHO recommends taking three blood pressure measurements. During data analysis, the average of the second and third readings is calculated. The participant must rest for one minute between each reading .

Heart rate measurement and recording should be done three times, along with blood pressure measurement and recording. The automatic tensiometer simultaneously presents the results.

The average of three measurements shall be calculated before the intervention and during the follow-up period.

24-hour urine collection: The urine sample will be collected in Plastic container: with capacity of three liters wide mouth BD Vacutainer, the second urine of the day until the first of the next morning. The sample shall be delivered on the agreed day for analysis.

The sodium in 24-hour urine excretion shall be estimated by selective ion electrode technology: the total sample shall be mixed, 200 μl shall be separated from the collected urine and diluted in 200 μl ml of urine diluent Urine thinner: (PN AV-BP0344D) company name and country of origin (if USA include state): Diluent used to analyze the urine sample in the electrolyte analyzer, (1:1 dilution). Select " urine mode" to analyze the sample. At the end, the results of the electrolytes Na, K and Cl will be reported on the screen. The result of the first measurement will be taken.They will be compared with the reference values, considering age and sex.

KontrolLab: Electrolyte Analyzer, KontroLab Analyzer is an in vitro diagnostic equipment manufactured with state-of-the-art technology, accurate, accurate and designed to be easy to use and maintain.

It is based on the properties of its transducers or sensors (electrodes) to be selective to a specific Ion in solution.

This is achieved thanks to the fact that the membranes of the Ion selective Electrodes develop a potential (with respect to a Reference electrode) proportional to the activity of the Ion in solution for which they are selective.

ISE Pack reagents: (PV AV-BP5186D) Include place of origin and company name: The package contains the following reagents for the calibration of sodium, potassium, chlorine, ionised calcium and lithium from the electrolyte analyser.

To obtain the value in mmol / 24 hours, it must be multiplied by the 24-hour sample volume of the patient, expressed in liters.

To blood pressure:

An automatic digital tensiometer validated according to the protocol for determining the sodium concentration, PAHO-WHO, 2010. It will be used marca OMRON: Model: HEM-7121.Distribuited by OMRON HEALTHCARE,INC.Illinois,U.S.A.

Intervention: They will be given recommendations for a low-sodium diet: Restriction of foods with high sodium content.

The duration time will be four weeks for assessment of BP and sodium excretion and consumption of foods high in salt; and at 24 weeks for the assessment of BP and consumption of foods high in salt.

Estimation of the consumption of fruits and vegetables,salt added to meals before and after meals and the consumption of industrialized products, at four and twenty-four weeks.

Physical activity and / or exercise will be assessed (type of exercise: aerobic or anaerobic and constancy: time 15 min, 30 min, 60 min, 120 min.

Questionnaire: identification of consumption fruits and vegetables, industrialized products, frequency, duration and type of exercise.

ELIGIBILITY:
Inclusion Criteria:

* Young men and women 18-40 years of age with diastolic blood pressure <90 and systolic blood pressure < 130.

Exclusion Criteria:

* Chronic non-hypertensive diseases
* Physical disability
* Subjects under treatment with diuretics
* Pregnant women, lactating or in their menstrual cycle
* High performance athletes

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 196 (Actual)
Dates: Start 2020-10-28 (Actual); Primary Completion 2023-05-09 (Actual); Study Completion 2023-05-09 (Actual)

PRIMARY OUTCOMES:
24-hour urine sodium excretion | up to 4 weeks
  mmol/l
blood pressure | up to 4 weeks
  mmHg

SECONDARY OUTCOMES:
24-hour urine potassium excretion | up to 4 weeks
  mmol/l
Physical activity | up to 4 weeks
  min

CONTACTS AND LOCATIONS:
Overall Officials: Arturo Jiménez-Cruz, Researcher, Study Director — University Autonomus of Baja California
Locations (1):
- Naysin Yaheko Pardo Buitimea, Tijuana, Estado de Baja California, Mexico

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD, all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: starting 1 month after publication
Access Criteria: by email

REFERENCES:
- [Result] Bakris G, Ali W, Parati G. ACC/AHA Versus ESC/ESH on Hypertension Guidelines: JACC Guideline Comparison. J Am Coll Cardiol. 2019 Jun 18;73(23):3018-3026. doi: 10.1016/j.jacc.2019.03.507. PMID 31196460
- [Result] Forrester T, Adeyemo A, Soarres-Wynter S, Sargent L, Bennett F, Wilks R, Luke A, Prewitt E, Kramer H, Cooper RS. A randomized trial on sodium reduction in two developing countries. J Hum Hypertens. 2005 Jan;19(1):55-60. doi: 10.1038/sj.jhh.1001782. PMID 15470483
- [Result] Stamler J, Chan Q, Daviglus ML, Dyer AR, Van Horn L, Garside DB, Miura K, Wu Y, Ueshima H, Zhao L, Elliott P; INTERMAP Research Group. Relation of Dietary Sodium (Salt) to Blood Pressure and Its Possible Modulation by Other Dietary Factors: The INTERMAP Study. Hypertension. 2018 Apr;71(4):631-637. doi: 10.1161/HYPERTENSIONAHA.117.09928. PMID 29507099
- [Result] Weinberger MH. Salt sensitivity is associated with an increased mortality in both normal and hypertensive humans. J Clin Hypertens (Greenwich). 2002 Jul-Aug;4(4):274-6. doi: 10.1111/j.1524-6175.2002.00924.x. PMID 12147930
- [Result] Drenjancevic-Peric I, Frisbee JC, Lombard JH. Skeletal muscle arteriolar reactivity in SS.BN13 consomic rats and Dahl salt-sensitive rats. Hypertension. 2003 May;41(5):1012-5. doi: 10.1161/01.HYP.0000067061.26899.3E. Epub 2003 Apr 7. PMID 12682080
- [Result] Drenjancevic-Peric I, Jelakovic B, Lombard JH, Kunert MP, Kibel A, Gros M. High-salt diet and hypertension: focus on the renin-angiotensin system. Kidney Blood Press Res. 2011;34(1):1-11. doi: 10.1159/000320387. Epub 2010 Nov 12. PMID 21071956
- [Result] Larsen SC, Angquist L, Sorensen TI, Heitmann BL. 24h urinary sodium excretion and subsequent change in weight, waist circumference and body composition. PLoS One. 2013 Jul 25;8(7):e69689. doi: 10.1371/journal.pone.0069689. Print 2013. PMID 23936079
- [Result] Fonseca-Alaniz MH, Brito LC, Borges-Silva CN, Takada J, Andreotti S, Lima FB. High dietary sodium intake increases white adipose tissue mass and plasma leptin in rats. Obesity (Silver Spring). 2007 Sep;15(9):2200-8. doi: 10.1038/oby.2007.261. PMID 17890487
- [Result] Smith-Spangler CM, Juusola JL, Enns EA, Owens DK, Garber AM. Population strategies to decrease sodium intake and the burden of cardiovascular disease: a cost-effectiveness analysis. Ann Intern Med. 2010 Apr 20;152(8):481-7, W170-3. doi: 10.7326/0003-4819-152-8-201004200-00212. Epub 2010 Mar 1. PMID 20194225
- [Result] Vedovato M, Lepore G, Coracina A, Dodesini AR, Jori E, Tiengo A, Del Prato S, Trevisan R. Effect of sodium intake on blood pressure and albuminuria in Type 2 diabetic patients: the role of insulin resistance. Diabetologia. 2004 Feb;47(2):300-3. doi: 10.1007/s00125-003-1303-5. Epub 2003 Dec 24. PMID 14704836
- [Result] Wilck N, Balogh A, Marko L, Bartolomaeus H, Muller DN. The role of sodium in modulating immune cell function. Nat Rev Nephrol. 2019 Sep;15(9):546-558. doi: 10.1038/s41581-019-0167-y. Epub 2019 Jun 25. PMID 31239546
- [Result] Strazzullo P, Cairella G, Campanozzi A, Carcea M, Galeone D, Galletti F, Giampaoli S, Iacoviello L, Scalfi L; GIRCSI Working Group. Population based strategy for dietary salt intake reduction: Italian initiatives in the European framework. Nutr Metab Cardiovasc Dis. 2012 Mar;22(3):161-6. doi: 10.1016/j.numecd.2011.10.004. Epub 2012 Feb 23. PMID 22364888
- [Result] Vega-Solano J, Blanco-Metzler A, Benavides-Aguilar KF, Arcand J. An Evaluation of the Sodium Content and Compliance with the National Sodium Reduction Targets among Packaged Foods Sold in Costa Rica in 2015 and 2018. Nutrients. 2019 Sep 15;11(9):2226. doi: 10.3390/nu11092226. PMID 31540146
- [Result] Manzel A, Muller DN, Hafler DA, Erdman SE, Linker RA, Kleinewietfeld M. Role of "Western diet" in inflammatory autoimmune diseases. Curr Allergy Asthma Rep. 2014 Jan;14(1):404. doi: 10.1007/s11882-013-0404-6. PMID 24338487
- [Result] Cavka A, Cosic A, Jukic I, Jelakovic B, Lombard JH, Phillips SA, Seric V, Mihaljevic I, Drenjancevic I. The role of cyclo-oxygenase-1 in high-salt diet-induced microvascular dysfunction in humans. J Physiol. 2015 Dec 15;593(24):5313-24. doi: 10.1113/JP271631. Epub 2015 Dec 7. PMID 26498129
- [Result] Meneton P, Jeunemaitre X, de Wardener HE, MacGregor GA. Links between dietary salt intake, renal salt handling, blood pressure, and cardiovascular diseases. Physiol Rev. 2005 Apr;85(2):679-715. doi: 10.1152/physrev.00056.2003. PMID 15788708
- [Result] Cook NR, Cutler JA, Obarzanek E, Buring JE, Rexrode KM, Kumanyika SK, Appel LJ, Whelton PK. Long term effects of dietary sodium reduction on cardiovascular disease outcomes: observational follow-up of the trials of hypertension prevention (TOHP). BMJ. 2007 Apr 28;334(7599):885-8. doi: 10.1136/bmj.39147.604896.55. Epub 2007 Apr 20. PMID 17449506
- [Result] Cook NR, Obarzanek E, Cutler JA, Buring JE, Rexrode KM, Kumanyika SK, Appel LJ, Whelton PK; Trials of Hypertension Prevention Collaborative Research Group. Joint effects of sodium and potassium intake on subsequent cardiovascular disease: the Trials of Hypertension Prevention follow-up study. Arch Intern Med. 2009 Jan 12;169(1):32-40. doi: 10.1001/archinternmed.2008.523. PMID 19139321
- [Result] Greaney JL, DuPont JJ, Lennon-Edwards SL, Sanders PW, Edwards DG, Farquhar WB. Dietary sodium loading impairs microvascular function independent of blood pressure in humans: role of oxidative stress. J Physiol. 2012 Nov 1;590(21):5519-28. doi: 10.1113/jphysiol.2012.236992. Epub 2012 Aug 20. PMID 22907057
- [Result] Rossi M, Carpi A, Galetta F, Franzoni F, Santoro G. The investigation of skin blood flowmotion: a new approach to study the microcirculatory impairment in vascular diseases? Biomed Pharmacother. 2006 Sep;60(8):437-42. doi: 10.1016/j.biopha.2006.07.012. Epub 2006 Aug 14. PMID 16935461
- [Result] Todd AS, Macginley RJ, Schollum JB, Williams SM, Sutherland WH, Mann JI, Walker RJ. Dietary sodium loading in normotensive healthy volunteers does not increase arterial vascular reactivity or blood pressure. Nephrology (Carlton). 2012 Mar;17(3):249-56. doi: 10.1111/j.1440-1797.2011.01550.x. PMID 22171802
- [Result] Gates PE, Tanaka H, Hiatt WR, Seals DR. Dietary sodium restriction rapidly improves large elastic artery compliance in older adults with systolic hypertension. Hypertension. 2004 Jul;44(1):35-41. doi: 10.1161/01.HYP.0000132767.74476.64. Epub 2004 Jun 1. PMID 15173128
- [Result] Mascioli S, Grimm R Jr, Launer C, Svendsen K, Flack J, Gonzalez N, Elmer P, Neaton J. Sodium chloride raises blood pressure in normotensive subjects. The study of sodium and blood pressure. Hypertension. 1991 Jan;17(1 Suppl):I21-6. doi: 10.1161/01.hyp.17.1_suppl.i21. PMID 1987006
- [Result] Caldeira D, Vaz-Carneiro A, Costa J. [What is the benefit of salt reduction on blood pressure? Assessment of the Cochrane Review: Effect of longer-term modest salt reduction on blood pressure. He FJ, Li J, Macgregor GA. Cochrane Database Syst Rev. 2013 Apr 30;4:CD004937]. Acta Med Port. 2013 Sep-Oct;26(5):490-2. Epub 2013 Oct 31. Portuguese. PMID 24192084
- [Result] Suckling RJ, He FJ, Markandu ND, MacGregor GA. Modest Salt Reduction Lowers Blood Pressure and Albumin Excretion in Impaired Glucose Tolerance and Type 2 Diabetes Mellitus: A Randomized Double-Blind Trial. Hypertension. 2016 Jun;67(6):1189-95. doi: 10.1161/HYPERTENSIONAHA.115.06637. PMID 27160199
- [Result] Chen J, Tian Y, Liao Y, Yang S, Li Z, He C, Tu D, Sun X. Salt-restriction-spoon improved the salt intake among residents in China. PLoS One. 2013 Nov 11;8(11):e78963. doi: 10.1371/journal.pone.0078963. eCollection 2013. PMID 24244395
- [Result] Aparicio A, Rodriguez-Rodriguez E, Cuadrado-Soto E, Navia B, Lopez-Sobaler AM, Ortega RM. Estimation of salt intake assessed by urinary excretion of sodium over 24 h in Spanish subjects aged 7-11 years. Eur J Nutr. 2017 Feb;56(1):171-178. doi: 10.1007/s00394-015-1067-y. Epub 2015 Oct 19. PMID 26482149
- [Result] Hoffmann IS, Cubeddu LX. Salt and the metabolic syndrome. Nutr Metab Cardiovasc Dis. 2009 Feb;19(2):123-8. doi: 10.1016/j.numecd.2008.02.011. Epub 2008 Jun 16. PMID 18556187
- [Result] Strazzullo P, D'Elia L, Kandala NB, Cappuccio FP. Salt intake, stroke, and cardiovascular disease: meta-analysis of prospective studies. BMJ. 2009 Nov 24;339:b4567. doi: 10.1136/bmj.b4567. PMID 19934192
- [Result] Kim J, Lim SY, Kim JH. Nutrient intake risk factors of osteoporosis in postmenopausal women. Asia Pac J Clin Nutr. 2008;17(2):270-5. PMID 18586647
- See also: Pan American Health Organization: PAHO/WHO — http://paho.org/hq/index.php?option=com_topics&view=article&id=221&Itemid=40878&lang=en